CLINICAL TRIAL: NCT06086821
Title: Clinical Relevance of Different Time of Periodontal Re-evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florence (Other)
Responsible Party: Principal Investigator, Luigi Barbato, Principal Investigator, University of Florence
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PerioTiming-1
Record Dates: First submitted 2023-10-10; First posted 2023-10-17 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Periodontal Diseases
Keywords: Periodontal Pocket; Periodontal treatment; Non-surgical periodontal treatment
MeSH Terms: conditions — Periodontal Diseases; Periodontal Pocket

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor does not know when Step 1 and 2 of periodontal treatment have been performed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3-Months (Active Comparator): Periodontal Re-evaluation performed three months after Step 2 have been completed.
  Interventions: Diagnostic Test: Periodontal Re-Evaluation
- 6-Months (Experimental): Periodontal Re-evaluation performed six months after Step 2 have been completed.
  Interventions: Diagnostic Test: Periodontal Re-Evaluation

INTERVENTIONS:
Diagnostic Test: Periodontal Re-Evaluation — Recording of the periodontal charting

SUMMARY:
Treatment of periodontitis follows an incremental step approach. The results after step 1 (Oral Hygiene Instruction and Professional Mechanical Plaque Removal) and 2 (subgingival instrumentation) are re-evaluated in order to understand whether the endpoints of therapy have been achieved.

The case reevaluation may be performed at different time intervals, ranging from 2 weeks to 6 months. The aim of this study is to compare two different timing of re-evaluation, in terms of clinical indexes (PPD reduction; Pocket closure) and patients' morbidity (number of further therapies needed).

DETAILED DESCRIPTION:
Treatment of periodontitis follows an incremental step approach in which the first step is aimed at modifying patient behavior with the goal of supragingival plaque reduction.

The second step is subgingival instrumentation, performed with different instruments and treatment timing and with or without additional therapies. However, in periodontitis patients, the complete removal of subgingival biofilm and calculus at teeth with deep probing depths (≥6 mm) or complex anatomical surfaces (root concavities, furcations, infra bony pockets) may be difficult, and hence, the endpoints of therapy may not be achieved, and further treatment should be implemented.

The third step of therapy is aimed at treating those areas of the dentition non-responding adequately to the second step of therapy (presence of pockets ≥4 mm with bleeding on probing or presence of deep periodontal pockets [≥5 mm]), with the purpose of gaining further access to subgingival instrumentation, or aiming at regenerating or resecting those lesions that add complexity in the management of periodontitis (intra-bony and furcation lesions).

Periodontal reevaluation is performed after step 2. The case reevaluation, executed after the completion of the first step of periodontal therapy, allows to assess the response to therapy, to specify the prognosis of the case and the possible need for further treatment and, consequently, to finalize and correct the case's periodontal treatment plan.

Many different time intervals, ranging from 2 weeks to 6 months, have been documented in periodontal literature to be the best time to perform reevaluation.

The decision on the timing of reevaluation is secondary to the expression of the clinical benefits of the first two steps of therapy. Classic studies show that the most significant changes occur during the first 3 months after instrumentation, with little change during the next 12 months.

Cugini studied the microbiological and clinical effect of subgingival instrumentation and found that most of the clinical improvements and microbial changes occurred during the first 3 months after SRP. In particular, the mean attachment level decreased significantly at 3 months and was maintained during the 12 months of the study. Other clinical parameters, such as mean pocket depth and the percentage of sites that bled on probing, showed marked improvement at 3 months after SRP, but also during the maintenance period.

Another study, in which 40 patients were randomized to Q-SRP or FMI showed that both therapies resulted in significant improvements in all clinical indices both at 6 weeks and 6 months. A continuous clinical improvement was seen for both treatment groups during the experimental period, which reached peak levels at 6 months.

A further study, that again compared two different approaches for sub-gingival instrumentation showed that the initial treatment phase resulted in ''pocket closure'' at a mean frequency of 58% for the FMD and 66% for the Q-SRP approach. Following re-treatment of the remaining pockets, the mean percentage of closed pockets increased to 74% for FMD and to 77% for Q-SRP.

A recent systematic review showed that, despite no differences exist on the mode of delivery of non-surgical therapy, at shallow sites (4-6 mm), a mean reduction of PD of 1.5 mm can be expected at 6/8 months, while at deeper sites (≥7 mm) the mean PD reduction was estimated at 2.6 mm. In addition, based on the results of 9 studies, the authors concluded that the proportion of closed pockets was estimated to be 57% and 74% at 3 and at 6 months, respectively.

Taking into account the overall patient, it becomes clear that the possibility of having an optimal effect (i.e. pocket closure) on a single site or a single tooth might have a minimum or a non-significant clinical effect on the overall treatment plan of a patient. The aim of this study is to compare two different timing of re-evaluation, in terms of clinical indexes (PPD reduction; Pocket closure) and patients' morbidity (number of further therapies needed).

Materials & Methods

This trial will be a single-blinded, randomized controlled clinical trial with a 6 months follow-up.

Following a screening examination including full-mouth probing and a radiographic evaluation, 40 patients will be recruited from the Department of Periodontology (AOU Careggi, Firenze).

Inclusion criteria:

Adults with a diagnosis of Generalized, stage III or stage IV periodontitis; At least 20 teeth present At least eight teeth must show probing pocket depths (PPD) of ≥5mm and bleeding on probing (BOP). At least two of these teeth must have a PPD of ≥7 mm and at additional two teeth, the pockets must measure ≥6 mm;

Exclusion criteria:

Patients receiving periodontal treatment in the past 12 months; Patients receiving antibiotics in the past 3 months; Known medical conditions that affects the progression of periodontitis or that affect the outcomes of periodontal therapy; Compromised medical conditions requiring prophylactic antibiotic coverage; and ongoing drug therapy that might affect the clinical signs and symptoms of periodontitis.

One examiner (an experienced periodontist, L. Barbato), who will be masked with respect to the treatment assignments, will retrieve all clinical recordings.

Full mouth clinical examination will be performed at baseline including clinical photos, full-mouth radiographs, along with a complete medical and dental history.

The enrolled subjects will be stratified according to smoking habits and randomly allocated to two different arms: (1) Subgingival instrumentation and re-evaluation at 3 months or (2) Subgingival instrumentation and re-evaluation at 6 months. To optimize the study design, step 1 periodontal therapy will be performed at the same time as step 2. To overcome possible bias due to different delivery timing of subgingival instrumentation, therapy will be delivered as a full mouth instrumentation or in two sessions one week apart. Therapy will be derived by post-graduate students with significant clinical experience in non-surgical therapy (post-graduate year 2 or 3). After baseline recordings and a detailed case presentation to the patient, the therapy will be delivered. The patients will be recalled monthly for re-enforcement of motivation and oral hygiene instruction and supra-gingival plaque removal. In the context of this appointments, no sub gingival re-instrumentation will be performed. At 3 months (group 1) and at 6 months (group 2) the same examiner will retrieve the re-evaluation periodontal chart.

According to recently published clinical guidelines for the treatment of stage III/IV of periodontitis, one of the authors (a periodontist with more than 10 years of experience, Cairo) will compile, for every clinical case, a complete corrective treatment plan, which may include non-surgical re-treatment, surgical conservative therapy, osseous resective therapy or regenerative therapy.

The definitive treatment plan will be drawn up and described for all those elements that have not achieved, after step 1 and 2 periodontal therapy, the therapeutic endpoints (no PPD≥5 mm and no PPD=4 mm with BOP).

Patient mean values will be calculated for the statistical analysis. The primary variable will be the number of teeth needing further therapies. Secondary variables will be PPD reduction, Pocket closure (i.e. no PPD≥5 mm and no PPD=4 mm with BOP), number of surgeries performed and also PROMs will be evaluated. A cost analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Adults with a diagnosis of Generalized, stage III or stage IV periodontitis;
* At least 20 teeth present
* At least eight teeth must show probing pocket depths (PPD) of ≥5mm and bleeding on probing (BOP). At least two of these teeth must have a PPD of ≥7 mm and at additional two teeth, the pockets must measure ≥6 mm;

Exclusion Criteria:

* Patients receiving periodontal treatment in the past 12 months;
* Patients receiving antibiotics in the past 3 months;
* Known medical conditions that affects the progression of periodontitis or that affect the outcomes of periodontal therapy;
* Compromised medical conditions requiring prophylactic antibiotic coverage; and ongoing drug therapy that might affect the clinical signs and symptoms of periodontitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Number of Teeth not reaching EoT (Endpoint of treatment) | 3 months after step 2 of periodontal treatment is completed
  Number of Teeth Needing further treatments
Number of Teeth not reaching EoT (Endpoint of treatment) | 6 months after step 2 of periodontal treatment is completed
  Number of Teeth Needing further treatments

CONTACTS AND LOCATIONS:
Locations (1):
- Università degli Studi di Firenze, Florence, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Castelluzzo W, Rupe C, Nieri M, di Martino M, Zini M, Sartori A, Tasco A, Spoleti F, Barbato L, Cairo F. Timing of Re-Evaluation After Periodontal Therapy: A Randomized Clinical Trial. J Periodontal Res. 2026 Feb 10. doi: 10.1111/jre.70086. Online ahead of print. PMID 41664833